CLINICAL TRIAL: NCT04487405
Title: A Multivariate Index Assay for Ovarian Cancer Risk Assessment in Women With Adnexal Mass and High-Risk Germline Variants
Acronym: OVAnex
Status: Terminated | Type: Observational
Why Stopped: cohort C looked at feasibility of genetics & protein to evaluate risk with a family hx of cancer or associated variant. Since few patients show these factors, this approach would not yield sufficient information to make inferences
Sponsor: Aspira Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 04-2019
Record Dates: First submitted 2020-07-10; First posted 2020-07-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Adnexal Mass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Symptomatic with adnexal mass
  Interventions: Device: OVAnex
- Group B: Asymptomatic with adnexal mass
  Interventions: Device: OVAnex
- Group C: Women with a predisposition in developing ovarian cancer due to a positive, pathogenic variant
  Interventions: Device: OVAnex

INTERVENTIONS:
Device: OVAnex — OVAnex is a multivarite index assay assessing ovarian cancer risk

SUMMARY:
The objective of this project is to validate the sensitivity, specificity, positive predictive value and negative predictive values of the AMRA blood test for assessing risk of cancer in women at high risk for ovarian cancer, due to the presence of a symptomatic adnexal mass.

ELIGIBILITY:
Inclusion Criteria:

* Female patient, 18 years of age or older diagnosed with an ovarian adnexal mass, or in follow-up due to the presence of BRCA1/2 and other germline DNA variants.
* Patient reviewed, understood, and provided the PI with written informed consent to allow blood specimen to be used for research and release of medical information.

Exclusion Criteria:

* Patient is less than 18 years of age
* Patient is not being treated in the U.S.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women with an ovarian adnexal mass, or in follow up due to the presence of BRCA1/2 and other germline DNA variants.
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
OVAnex | 12 months
  OVAnex is a multivariate index assay assessing ovarian cancer risk. The Ovanex MIA uses seven biomarkers with a stepwise algorithm to generate a risk score which ranges from 0 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Pappas, PhD, Principal Investigator — Aspira Women's Health
Locations (9):
- United States (9):
  - Women's Health Arizona, Chandler, Arizona
  - Altus Research, Lake Worth, Florida
  - MidTown OBGYN, Columbus, Georgia
  - Premier OBGYN of Minnesota, Eden Prairie, Minnesota
  - Square Care Health, New Hyde Park, New York
  - Northwell Health, New Hyde Park, New York
  - Seven Hills Clinical Research Group, Cincinnati, Ohio
  - May Grant OB/GYN, Lancaster, Pennsylvania
  - Hill Country OBGYN Associates, Austin, Texas

IPD SHARING:
Plan to Share IPD: No